CLINICAL TRIAL: NCT00083018
Title: Evaluation Of The Role Of Nipple Aspiration, Ductal Lavage And Duct Endoscopy At The Time Of Surgery In Patients With Breast Cancer
Brief Title: Nipple Aspiration, Ductal Lavage, and Duct Endoscopy For Diagnostic Assessment in Women Undergoing Surgery for Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000361760; RMNHS-2283; EU-20353
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2005-12

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IA breast cancer; stage IB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cytogenetic Analysis; Immunohistochemistry

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: proteomic profiling
Other: cytology specimen collection procedure
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: breast duct lavage

SUMMARY:
RATIONALE: Diagnostic procedures, such as nipple aspiration, ductal lavage, and breast duct endoscopy, may help doctors detect and assess breast cancer cells early and plan more effective treatment.

PURPOSE: This phase II trial is studying how well nipple aspiration, ductal lavage, and duct endoscopy work in assessing cancer cells in women who are undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Correlate the cell yield and morphology findings from ductal lavage with duct endoscopy findings and surgical pathology findings in women with breast cancer.
* Determine the sensitivity and specificity of nipple aspiration, ductal lavage, and duct endoscopy in detecting established breast cancer in these patients.

Secondary

* Compare the intraduct environment of cancer-involved ducts in the affected breast vs the ductal systems in the contralateral breast of these patients.
* Perform immunohistochemical analysis (including estrogen receptor, progesterone receptor, HER2-neu receptor, epidermal growth factor receptor, p53, and proliferation marker expression) for markers potentially associated with breast cancer in these patients.
* Determine potential molecular markers of malignancy by gene methylation, gene expression, and proteomics in these patients.
* Compare the biochemistry and protein analysis of the intraductal fluid vs serum analysis in these patients.

OUTLINE: Patients undergo nipple aspiration, ductal lavage, and duct endoscopy under general anesthesia immediately before breast surgery. Fluid and tissue obtained are examined for tumor markers by immunohistochemistry. Candidate genes are analyzed by gene methylation, gene expression arrays, and proteomic profiling.

Patients are followed at 24 hours and at 1 week.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* No metastatic disease
* No inflammatory breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No active infection or inflammation in the breast under study
* No known allergy to eutectic mixture of local anesthetics (EMLA®) cream or lidocaine
* No severe illness
* Not unconscious
* No mental illness or handicap
* No nursing within the past 12 months
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior breast implantation on side of proposed lavage
* No prior subareolar (e.g., papilloma resections, biopsies, or fine needle aspirations) or other surgery that may disrupt the ductal systems within 2 cm of the nipple

  * Biopsies and fine-needle aspirations > 2 cm from the nipple are allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-09

PRIMARY OUTCOMES:
Correlation of cell yields and morphology in ductal lavage with duct endoscopy appearances and findings
Sensitivity and specificity of ductal lavage with or without ductoscopy in detecting atypical cells
Comparison of cell yields vs final surgical pathology of the operative specimens

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gui, MD, MS, FRCS(Edin), FRCS(Eng), Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - London, London, England, United Kingdom